CLINICAL TRIAL: NCT00401934
Title: Protective Immunity to Human Cholera in Bangladesh
Brief Title: Immunity to Human Cholera in Bangladesh
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 06-0045
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2011-08

CONDITIONS: Cholera
Keywords: cholera, Vibrio cholerae, diarrhea, Bangladesh, children
MeSH Terms: conditions — Cholera; Diarrhea

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Cholera is a severe diarrhea illness caused by bacteria. The purpose of this study is to better understand how the immune systems of people in Dhaka, Bangladesh, fight infection with cholera. Understanding immune responses that influence the outcome of infection with cholera can assist in the development of more effective cholera vaccines. The International Center for Diarrheal Diseases Research, Bangladesh (ICDDR,B) will enroll in this study 75 patients with acute cholera and 250 of their household contacts. Individuals ages 2-60 years are eligible. Study participation will last 1 year for cholera patients and 30 days for household contacts. Participants will come to the ICDDR,B for 3 (household contacts) or 4 (cholera patients) study visits, and field workers will visit them at home at other times. For all participants, blood samples will be taken at each of the ICDDR,B visits. Household contacts will have rectal swabs taken at 2 ICDDR visits and during field worker visits.

DETAILED DESCRIPTION:
The purpose of this study is to investigate protective immunity to human cholera in Dhaka, Bangladesh. Immune responses to Vibrio cholerae are poorly understood and have not been extensively studied in an endemic setting such as Bangladesh. Understanding systemic and mucosal immune responses that influence the outcome of infection with V cholerae can assist in the development of more effective cholera vaccines. Identifying host factors, such as human genetic variations or nutritional status, that affect the outcome of infection with V cholerae can lead to an improved understanding of disease pathogenesis and better treatment modalities. One of the likely key determinants of protection following either natural cholera or vaccination is the duration of immune responses to key antigens, particularly at the mucosal surface. This study proposes to assess the duration of immune responses in a group of 75 cholera study participants over the course of 1 year of follow-up and to correlate baseline immune responses in 250 household contacts of the index patients, with protection from disease over the subsequent 30 days. The researchers will assess the duration of immunity in serum to known cholera virulence factors, including the serum vibriocidal antibody and antibodies specific for LPS, cholera toxin, B subunit (CtxB), and TcpA. The researchers will also measure antigen-specific memory B cells circulating in human blood, which has previously been used to examine the longevity of B cell immunologic memory following various infections and vaccinations. The objectives of this study are to determine genes and proteins expressed by V. cholerae during human infection; determine which V. cholerae proteins are immunogenic during human cholera infection in Bangladesh; assess the duration of immune responses to V. cholerae antigens following an episode of cholera; determine which anti-V. cholerae immune responses are protective on exposure to cholera in household contacts; and evaluate selected host factors that influence the development of immune responses following cholera, or susceptibility to symptomatic cholera following exposure in household contacts. A total of 325 study participants (75 index patients with acute cholera and 250 of their household contacts) will be enrolled. Index study participants will be recruited from among patients presenting with acute cholera to the International Center for Diarrheal Diseases Research, Bangladesh (ICDDR,B) hospital in Dhaka, Bangladesh. Any individual with acute cholera between the ages of 2 to 60 years, inclusive, without a severe complicating illness, and any household contact of the cholera patients between the ages of 2 and 60 years, inclusive, is eligible for enrollment in this study. The length of participation for each study participant will be 1 year for acute cholera index patients and 30 days for their household contacts. For cholera patients, study physicians will perform an initial assessment and collect blood at various time points over 1 year. Study participants (cases and household contacts) will come to the ICDDR,B for blood collection. On Study Days 3 through 6 and 8 through 10, a trained field worker will visit the household contacts to collect information about symptoms and treatment of diarrhea and to obtain rectal swab samples. Household contacts will come to the ICDDR,B on Days 2 or 3, and 7 (range 6-9) for a questionnaire, rectal swab, and blood drawing. Questionnaires will be filled out upon enrollment and at each study visit.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Men or women age 2 to 60 years, inclusive.
* Provision of informed consent for enrollment in study by patient/parent or guardian, as well as verbal assent for children age 7 to 17 years, inclusive.
* Expressed interest and availability to fulfill the study requirements (index patients for up to 1 year; household contacts up to 30 days).

Index Patients:

- Any individual with cholera enrolled in the surveillance system at the International Centre for Diarrhoeal Diseases Research, Bangladesh (ICDDR,B).

Household Contacts:

- Any household contact of the index patient (defined as sharing the same cooking pot for longer than 3 days before the index patient presented to the ICDDR,B).

There is no upper limit on the number of household members that can enroll from a single household.

Exclusion Criteria:

* Clinically apparent severe comorbid condition (meningitis, encephalitis, coma, respiratory distress).
* Concurrent enrollment in an unrelated interventional study.
* For household contacts, living in the same place with an index patient for 3 or fewer days before the index patient presented to the International Centre for Diarrhoeal Diseases Research, Bangladesh.

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400
Dates: Start 2006-12-11; Primary Completion 2012-01-04 (Actual); Study Completion 2012-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrhoeal Disease Research, Dhaka, Bangladesh